CLINICAL TRIAL: NCT02972983
Title: Daptomycin as Adjunctive Therapy for Staphylococcus Aureus Bacteremia
Acronym: DASH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Todd Lee, Doctor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-2666
Record Dates: First submitted 2016-11-21; First posted 2016-11-25 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Methicillin Susceptible Staphylococcus Aureus Septicemia; Bacteremia
Keywords: Staphylococcus aureus; Bacteremia; Daptomycin
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections | interventions — Daptomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 51 patients receiving a daily placebo infusion for five days on top of standard of care treatment for methicillin-sensitive Staphylococcus aureus (MSSA) bacteremia
  Interventions: Other: Placebo
- Daptomycin (Experimental): 51 patients receiving daily daptomycin infusion for five days on top of standard of care treatment for MSSA bacteremia
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Adjuvant therapy for up to five days
  Other Names: Cubicin
  Arms: Daptomycin
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of our study is to examine the effects of a second antibiotic, daptomycin, in combination with a beta lactam antibiotic on treating bloodstream infection caused by methicillin-susceptible S. aureus.

DETAILED DESCRIPTION:
When patients have a blood infection with methicillin-susceptible S. aureus, they will all be treated with the usual standard of care, including abeta-lactam antibiotic, have their blood tested daily for the presence of the infection until they test negative, as well as an ultrasound of the heart to rule out an infection of the heart valves, as well as have any catheters removed (if possible) to ensure adequate control of the infection.

This study involves adding a second antibiotic, daptomycin, to the treatment regimen of half of the patients enrolled in this study. Daptomycin is approved by Health Canada for treating blood infections due to Staphylococcus aureus. It is currently not used in combination with a beta-lactam for these infections because there is insufficient evidence of benefit to justify the cost.

The study participants will receive an additional daily iv therapy which will consist of either daptomycin or a placebo for a total of five days while admitted to the hospital. During this time, the participants will continue to have their blood drawn to assess for the presence of bacteria. The participants' liver and muscle enzymes will also be measured on the first and fifth day of therapy to test for potential side effects of the daptomycin.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a methicillin susceptible Staphylococcus aureus bacteremia.

Exclusion Criteria:

* Underlying terminal illness
* Significant contraindication to beta-lactam therapy (i.e. severe allergy, severe adverse drug reaction)
* Expected death before 5 days
* Microbiologically confirmed need for concomitant VANCOMYCIN or DAPTOMYCIN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Blood culture clearance | 5 days
  Time between first positive and first negative blood culture

SECONDARY OUTCOMES:
Mortality | 30 days
  Death from all causes (yes/no)
Adverse Reactions | 5 days
  Daptomycin adverse reactions
Intensive care admission | 30 days
  Admission to the intensive care unit (yes/no)
Metastatic infection | 30 days
  The development of a new deep seated infection (e.g. osteomyelitis, abscess, endocarditis) not present at time of initial bacteremia
Recurrent infection | 30 days
  The presence of a new positive blood culture occurring after the first negative culture and within 30 days of the initial positive

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre (Royal Victoria Hospital, Montreal Neurological Hospital, and Montreal General Hospital), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We will make this available under the right conditions including the appropriate data sharing agreements and ethics applications under Quebec law.

REFERENCES:
- [Background] Cheng MP, Lawandi A, Butler-Laporte G, Paquette K, Lee TC. Daptomycin versus placebo as an adjunct to beta-lactam therapy in the treatment of Staphylococcus aureus bacteremia: study protocol for a randomized controlled trial. Trials. 2018 May 29;19(1):297. doi: 10.1186/s13063-018-2668-6. PMID 29843781
- [Background] Cheng MP, Lawandi A, Butler-Laporte G, De l'Etoile-Morel S, Paquette K, Lee TC. Adjunctive Daptomycin in the Treatment of Methicillin-susceptible Staphylococcus aureus Bacteremia: A Randomized, Controlled Trial. Clin Infect Dis. 2021 May 4;72(9):e196-e203. doi: 10.1093/cid/ciaa1000. PMID 32667982